CLINICAL TRIAL: NCT00301288
Title: A Retrospective Study of Toxicity and Outcome of High Dose Chemotherapy With Autologous Stem Cell Transplant in Patients With Non-Hodgkin Lymphoma (NHL).
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: 2657
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Autologous stem cell transplant

SUMMARY:
Patients with aggressive Non-Hodgkin-lymphoma treated at first diagnosis with chemotherapy alone or combined chemo-radiotherapy can achieve high response rates. However, patients with relapsed lymphoma still have a poor prognosis. High dose chemotherapy (HDCT) followed by autologous stem cell transplantation (ASCT) is the treatment of choice for these patients. An ASCT allows patients to receive much higher doses of chemotherapy than usual, to improve the chances of curing the disease. The high-dose of chemotherapy destroys the cells in the patients bone marrow and then the patients own cells from either the bone marrow or peripheral blood are used to rescue the patient from intensive treatment. High-dose chemotherapy with autologous stem cell (either bone marrow or peripheral blood) transplantation is used in the treatment of Intermediate/High grade NHL with poor risk disease and in second remission at the Royal Marsden Hospital.

The purpose of the present analysis is to determine independent prognostic factors correlated with the long-term outcome of patients with NHL who received an ASCT between January 1991 and June 2005. Accrual of eligible patients currently under follow-up will be performed in clinic at the time of next appointment. All patients accrued will give informed consent to participate in the study for retrospective case note review, after discussion with a study investigator and after receiving a study information sheet. The results of the analysis will be published in a peer-reviewed medical journal. This will include patients treated at the royal Marsden Hospital only.

ELIGIBILITY:
Inclusion Criteria:

- a) Age over 18 b) Patients with Non-Hodgkin's Lymphoma who have received an autologous stem cell transplant in the past.

c) Informed written consent

Exclusion Criteria:

* a) Medical or psychiatric conditions that compromise the patient's ability to give informed consent b) HIV positive or AIDS related lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 152 participants with Non-Hodgkin's Lymphoma who have received an autologous stem cell trandplant in the past and have written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 152

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS trust, Sutton, Surrey, United Kingdom